CLINICAL TRIAL: NCT02438878
Title: Supporting Baby Behavior Through Pediatric Offices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 687861; WIC NEI-12-TX (Other: UC Davis)
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Infant Behavior; Feeding Behavior; Breastfeeding; Pediatric Obesity
MeSH Terms: conditions — Infant Behavior; Feeding Behavior; Breast Feeding; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baby Behavior (Experimental): The intervention is comprised of 2 components: HCP and medical staff training and participant education. The trainings will be video-based and aim to build providers' knowledge and skills to support parents' recognition and understanding of common healthy infant behaviors that may be misinterpreted by parents. The intervention does not include any specific recommendations for infant feeding, nor does it include any information related to the assessment, diagnosis or treatment for any medical condition.
  After completion of the intervention trainings, health care providers and medical staff will be asked to use what they learned with the mothers of infants in their care. Short handouts for mothers will be provided as tools to reinforce the verbal education. All educational materials will be focused only on supporting parents' abilities to recognize and understand common, healthy infant behaviors.
  Interventions: Behavioral: Baby Behavior
- Control (No Intervention): The control arm will continue with standard well-baby visit practices during the intervention period and will be offered the option to complete the Baby Behavior online trainings for continuing education credits.

INTERVENTIONS:
Behavioral: Baby Behavior
  Arms: Baby Behavior

SUMMARY:
The primary objective of this project is to evaluate the impact on infant growth and infant-feeding practices of a low-cost series of video trainings and tools targeted to medical staff and designed to support ongoing Baby Behavior education of WIC participants.

DETAILED DESCRIPTION:
The primary objective of this project is to evaluate the impact on infant growth and infant-feeding practices of a low-cost series of video trainings and tools targeted to medical staff and designed to support ongoing Baby Behavior education of WIC participants. The intervention, currently used in all California WIC agencies, teaches caregivers to recognize and understand healthy infant behaviors such as the range of infant cues and common patterns for sleep and crying. This project will also evaluate the acceptance, knowledge transfer, and use of the tools by health care providers and medical staff. It is expected that trained staff will be prepared to share Baby Behavior messages with their patients and that the information will be delivered quickly and easily during well-baby visits.

ELIGIBILITY:
Inclusion Criteria:

* Will attend a participating pediatric clinic for her well-baby visits
* Primiparous, singleton pregnancy
* Currently enrolled in WIC
* At least 18 years of age
* Speaks and reads English or Spanish
* Has a telephone and access to the internet
* Plans to stay in the area for 6 months after birth of infant
* Abstained from smoking during pregnancy

Exclusion criteria:

* Gave birth before 37 weeks gestation
* She and/or her infant has health condition(s) or known health risks that contraindicate breastfeeding
* She and/or her infant has health condition(s) or known health risks that impact infant growth and development

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2017-02-16 (Actual)

PRIMARY OUTCOMES:
Weight-for-length growth trajectory | Up to 6 months postpartum
  Weight-for-length Z scores calculated using the WHO Multicenter Growth Standards

SECONDARY OUTCOMES:
Infant feeding practices | 1 week, 2 weeks, 2 months, 4 months, and 6 months postpartum
  Breastfeeding duration and exclusivity, introduction of non-breast milk foods and fluids, use of sugary beverages, and intake of formula and select complementary foods
Maternal depressive symptoms | 2 weeks and 6 months postpartum
  Edinburgh Postnatal Depression Scale
Maternal self-efficacy | 1 week, 2 months, and 6 months postpartum
  Perceived Maternal Parenting Self-Efficacy
Maternal perceived stress | 1 week, 2 months, and 6 months postpartum
  Perceived Stress Scale Short-Form
Infant sleep patterns | 2 months and 6 months postpartum
  Brief Infant Sleep Questionnaire
Infant development | 2 months, 4 months, and 6 months postpartum
  Ages and Stages Questionnaire
Infant eating behavior | 4 months postpartum
  Baby Eating Behavior Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jane Heinig, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Davis, California, United States